CLINICAL TRIAL: NCT05769790
Title: Droplet-digital PCR for the Detection of Circulating Cell-free DNA in Patients With Cystic Echinococcosis: an Exploratory Study
Acronym: Echino_ddPCR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-02
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Cystic Echinococcosis
MeSH Terms: conditions — Echinococcosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ddPCR — The search for cfDNA will be performed using assays available in the literature for the search for E. granulosus cfDNA developed for PCR analysis in biological samples, targeting EgG1 Hae III repeat region, cox1 and nad1 (Zhao et al 2021). Appropriate controls (synthetic sequences and Parasitic reference DNA, provided by the Echinococcosis Reference Center of the Istituto Superiore di Sanità, Rome) will be included in each experiment.

SUMMARY:
It is an experimental study, multicentre, non-profit, whose aim is to preliminarily evaluate the sensitivity of ddPCR for the detection of cfDNA in the diagnosis of cystic echinococcosis and to generate data for its potential use also for the discrimination of the presence of infection with active/inactive cysts and the post-therapy follow-up.

DETAILED DESCRIPTION:
It is an experimental study, multicentre, non-profit, whose aim is to preliminarily evaluate the sensitivity of ddPCR for the detection of cfDNA in the diagnosis of cystic echinococcosis and to generate data for its potential also use for discrimination of the presence of infection with active/inactive cysts and follow-up aftercare, to be explored in subsequent studies. For this purpose, the plasma of adult patients with untreated hepatic cystic echinococcosis will be analysed.

The analyzes will be carried out on samples of patients who have already had a definitive diagnosis of cystic echinococcosis, and therefore the results of the study analyzes will have no influence on the diagnosis and clinical management of the patient, which, therefore, will not be informed of the result of the analyzes relating to his/her sample.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years;
2. definite diagnosis of hepatic cystic echinococcosis, ascertained on the basis of the presence of at least one liver cyst with pathognomonic signs on ultrasound examination or the presence of at least one liver cyst without clearly visible pathognomonic signs but presence of positive serology with at least two validated commercial tests or western blot (LDBIO Diagnostics, Lyon, France) positive for anti-Echinococcus antibodies (WHO-IWGE diagnostic criteria, Brunetti et al 2010);
3. no prior therapy for cystic echinococcosis reported;
4. willingness to participate in the study by signing the Informed Consent form.

Exclusion Criteria:

1. age < 18 years;
2. unconfirmed diagnosis of cystic echinococcosis; Echino_ddPCR version 1.1 of 02/14/2022
3. presence of echinococcal cysts only in extra-hepatic localization;
4. history of treatment for cystic echinococcosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
ddPCR sensitivity | 6 months
  Number of subjects with E. granulosus s.l. cfDNA detected by ddPCR in plasma, in relation to the total number of subjects with certain diagnosis untreated hepatic cystic echinococcosis

SECONDARY OUTCOMES:
ddPCR sensitivity by cyst stage | 6 months
  Number of subjects with cfDNA of E. granulosus s.l. detected by ddPCR in plasma, in ratio to the total number of subjects with certain diagnosis of hepatic cystic echinococcosis not treated divided by the presence of active and inactive cysts.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Fondazione Policlinico San Matteo, Pavia, PV
  - IRCCS Sacro Cuore Don Calabria hospital, Negrar, Verona